CLINICAL TRIAL: NCT06656845
Title: Feasibility of a Self-management App for People With Knee Osteoarthritis (OA-AID Feasibility Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Anne Therese Tveter, Professor, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 786516
Record Dates: First submitted 2024-10-08; First posted 2024-10-24 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthristis
Keywords: Osteoarthritis; E-health; Remote care; Feasibility
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- To determine the feasibility of a patient self-management app in patients with knee osteoarthritis (Experimental): The intended purpose of the app (Genus) is to provide information on osteoarthritis and recommended treatment for people with knee OA.
  Interventions: Device: Genus, a self-management app for patients with knee osteoarthritis

INTERVENTIONS:
Device: Genus, a self-management app for patients with knee osteoarthritis — The self-management app (Genus) will include weekly reminders with information videos on knee osteoarthritis and treatment options, exercise videos, quizzes, questionnaires, and a platform for remote monitoring by health professionals.

SUMMARY:
In this feasibility trial, an 8-week digital intervention including remote monitoring in patients with knee osteoarthritis (OA) will be tested. The app will provide information on osteoarthritis and recommended treatment for people with knee OA.

DETAILED DESCRIPTION:
In this feasibility study various outcome measures will be assessed to determine whether the app (Genus) is viable, practical, and useful.

The study will test the feasibility of an 8-week digital intervention including remote monitoring prior to consultation in specialist healthcare. The app consist of information on osteoarthritis and recommended treatment for people with knee OA. A total of 20 patients referred to Diakonhjemmet Hospital due to knee OA will be recruited to the study. The study will include assessments of technical, operational, clinical, and trial aspects of feasibility. Data will be collected through digital questionnaires (through the app or Nettskjema), through interviews and from medical records. Primary outcome is the feasibility of the app after 8 weeks. Additionally, the feasibility of the study process until consultation in specialist healthcare will be assessed.

The aim of the app is to improve patients' health literacy and enhance the shared decision-making process between patient and healthcare provider at the consultation in specialist healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Men and women =>50 years of age
* Referred to specialist healthcare for knee OA management

Exclusion Criteria:

* Received joint replacement or are under consideration for revision in the referred joint
* Have uncontrolled serious comorbidities
* Have cognitive dysfunction
* Are seeking care for trauma conditions or psoriatic/rheumatoid arthritis
* Unable to understand Norwegian
* Do not have a smartphone

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Desirable feasibility level | Through the 8 weeks intervention period
  Acceptable overall feasibility of the app with ≥70% of the secondary endpoints indicating feasibility

SECONDARY OUTCOMES:
Patient-reported software usability | At 8 weeks
  Considered feasible if the System Usability Scale score ≥68 on a 0-100 scale, 100= best score).
Patient-reported experiences and perceived benefits | At 8 weeks
  Experiences and perceived benefits collected in semi-structured interview
Patient-reported satisfaction with the app | At 8 weeks
  Measured by a numeric rating scale (NRS) 0-10, higher scores indicate better outcome. Acceptable feasibility 70% with score ≥5
Integration of workflow for health professionals | At baseline
  Measured by registering time of time use: acceptable feasibility if <30 minutes is spent on screening and enrolling (consent, baseline questionnaire, and downloading).
Time use in the intervention period | Through the 8 weeks intervention period
  Acceptable feasibility if <10 minutes are spent in max 1/3 of the patients
Primary clinical outcome | At baseline and at study completion (approx. 3 months after inclusion)
  Available data on total score in the Knee Osteoarthritis Knowledge Scale (KOAKS, scored on a scale from 11-55) at baseline and after intervention for ≥80% of patients.
Patient satisfaction with the intervention at 8 weeks | At 8 weeks
  Considered feasible if 70% with score ≥5 on a numeric rating scale (NRS) 0-10 on patient satisfaction with intervention.
Other patient reported outcomes | At 8 weeks
  Available data at 8 weeks for ≥80% of the patients
Recruitment rate | At baseline
  Acceptable recruitment rate is ≥50% of eligible patients
Patient dropout | At 8 weeks
  Number of patients that withdraw from the study. Acceptable withdrawal rate is ≤20% of included patients.
Trial logistics as assessed through interviews | At study completion (approx. 3 months after inclusion)
  Acceptable overall trial logistics as evaluated by the study group.
Patients' app use | Through study completion (approx. 3 months after inclusion)
  Acceptable app use includes that ≥50% of the patients watch ≥80% of the videos (16 videos), ≥50% of the patients has exercised1 or more days, ≥50% have completed at least 1 quiz.
Potential risk and challenges as assessed through interviews | At study completion (approx. 3 months after inclusion)
  Identify potential risk and challenges that could hinder a successful clinical evaluation of the app in a large randomised, controlled trial: Acceptable overall potential risk and challenges as evaluated by the study group at end of study.
Software performance and functionality | Through study completion (approx. 3 months after inclusion)
  Acceptable number of errors (≤3 errors per patient) in the performance and functionality experienced by the patients and project group members
Other patient reported outcomes | Through study completion (approx. 3 months after inclusion)
  Available data on other patient reported outcomes at pre- and post-consultation questionnaires for ≥80% of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Anne Therese Tveter, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No